CLINICAL TRIAL: NCT00491101
Title: Valuation of Quality of Life in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Iwona Stelmach MD, PhD, Prof, Department of Pediatrics and Allergy, Medical University of Lodz, Poland.
Other Study IDs: RNN-82-07-KE
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2008-12

CONDITIONS: Asthma
Keywords: Asthma Control; Quality of Life; Children; Polish Version of PAQLQ(S) by Juniper
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Children with asthma, both genders, from 7-18 years old.
  Interventions: Other: Polish Version of PAQLQ(S) by Juniper; Other: spirometry

INTERVENTIONS:
Other: Polish Version of PAQLQ(S) by Juniper — Polish Version of PAQLQ(S) by Juniper
Other: spirometry — spirometry

SUMMARY:
The aim of the study is valuation of quality of life (QL) in children with asthma and analysis of the factors that can have influence on it. The clinical problems included into the aim are to evaluate:

* the correlation between the QL and asthma control
* the utility of the Polish Version of PAQLQ(S) by Juniper, especially the understanding of each question and it's answers The results of this study can be very helpful in the future in developing a questionnaires to use in Polish Primary Care, according to which the investigators would be able to see whether the asthma in our patients is being well controlled.

DETAILED DESCRIPTION:
Quality of Life in people with asthma is strictly relevant with the correct treatment of the disease, that is why the correct screening of patient's quality of life, especially in children, is so important.

Exploring the quality of life (QL), we use different types of questionnaires to obtain a quantitative result, which we can interpret using a compatible key for it. Pediatric Asthma Quality of Life Questionnaire with Standardized Activities (PAQLQ(S)) by Juniper is a reliable measure of the influence of asthma on QL in children. The Polish Version of the questionnaire is a strict translation of the english one, however it is not completely validated, which in practice can evince in difficulties in understanding the meaning of the applied questions, probably because of the difference in the habits of both populations.

The aim of the study is valuation of quality of life (QL) in children with asthma and analysis of the factors that can have influence on it. The clinical problems included into the aim are to evaluate:

* the correlation between the QL and asthma control
* the utility of the Polish Version of PAQLQ(S) by Juniper, especially the understanding of each question and it's answers The results of this study can be very helpful in the future in developing a questionnaires to use in Polish Primary Care, according to which we would be able to see whether the asthma in our patients is being well controlled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Asthma
* Asthma treatment at least 6 months before enrollment
* Must be able to do spirometry

Exclusion Criteria:

* Children during the introductory period of the specific immunotherapy
* Other protracted diseases

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with asthma.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Daniela Gjurow, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Poland, Lodz, Poland